CLINICAL TRIAL: NCT04093258
Title: Comparison of Two Silicone Hydrogel Multifocal Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6344
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Results first posted 2021-02-16 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test/Control (Experimental): Eligible subjects between 40-70 years of age who are habitual soft contact lens wearers and hyperopic or myopic and have presbyopia will be randomized to one of two sequences (Test/Control or Control/Test) with a 4-10 day washout period in between each fitting.
  Interventions: Device: Dailies Total 1® Multifocal Contact Lenses; Device: Air Optix® Multifocal Contact Lenses Plus HydraGlyde®
- Control/Test (Experimental): Eligible subjects between 40-70 years of age who are habitual soft contact lens wearers and hyperopic or myopic and have presbyopia will be randomized to one of two sequences (Test/Control or Control/Test) with a 4-10 day washout period in between each fitting.
  Interventions: Device: Dailies Total 1® Multifocal Contact Lenses; Device: Air Optix® Multifocal Contact Lenses Plus HydraGlyde®

INTERVENTIONS:
Device: Dailies Total 1® Multifocal Contact Lenses — TEST
Device: Air Optix® Multifocal Contact Lenses Plus HydraGlyde® — CONTROL

SUMMARY:
This is a single-masked, randomized-controlled, dispensing clinical trial. A total of approximately 40 eligible hyperopic and myopic subjects will be targeted to complete the study. The subjects will be fit in the first study lens and worn for a total of 8-12 days following a 7±3 day wash-out period. The procedures will be repeated for the 2nd lens.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all the following criteria to be enrolled in the study:

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. The subject must be between 40 and 70 years of age (inclusive).
  4. The subject's distance spherical equivalent refraction must be in the range of +1.25 D to +3.75 D or -1.25 D to -4.00 D in each eye.
  5. The subject's refractive cylinder must be ≤0.75 D in each eye.
  6. The subject's ADD power must be in the range of +0.75 D to +2.50 D.
  7. The subject must have best corrected visual acuity of 20/20-3 or better in each eye.
  8. Subjects must own a wearable pair of spectacles if required for their distance vision.
  9. The subject must be an adapted soft contact lens wearer in both eyes (i.e. worn lenses a minimum of 2 days per week for at least 8 hours per wear day, for 1 month of more duration).
  10. The subject must either already be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".

      Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating.
  2. Any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.
  3. Any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
  4. Clinically significant (Grade 3 or 4) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
  5. Entropion, ectropion, extrusions, chalazia, recurrent styes, dry eye, glaucoma, history of recurrent corneal erosions.
  6. Any previous, or planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, lid procedures, dacryocystorhinostomy, cataract surgery, retinal surgery, etc.).
  7. A history of amblyopia, strabismus or binocular vision abnormality.
  8. Any current ocular infection or inflammation.
  9. Any current ocular abnormality that may interfere with contact lens wear.
  10. Use of any of the following oral medications within 1 week prior to enrollment: oral retinoid isotretinoin (e.g. Accutane), oral tetracyclines, topical scopolamine, oral antihistamines (e.g., Chlor-Trimeton, and Benadryl), systemic steroids.
  11. Use of any ocular medication, with the exception of rewetting drops.
  12. History of herpetic keratitis.
  13. Participation in any contact lens or lens care product clinical trial within 7 days prior to study enrollment.
  14. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
  15. Any known hypersensitivity or allergic reaction to OPTI-FREE® Puremoist® multipurpose care solution, sodium fluorescein or single-use preservative free rewetting drop solution.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Visual Eyes, Roswell, Georgia
  - ProCare Vision Centers, Granville, Ohio
  - Optometry Group, LLC, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total, 42 subjects were enrolled in this study; of which, 41 were randomly assigned into 2 sequences while, 1 subject failed to meet all eligibility criteria. Of the total assigned subjects, 40 subjects completed the study while, 1 subject was discontinued from the study.
Groups:
- Test/Control: Subjects randomized to this sequence received the Test lens during the first period and then received the Control lens during the second period.
- Control/Test: Subjects randomized to this sequence received the Control lens during the first period and then received the Test lens during the second period.
Period: Period 1
Arm/Group | Test/Control | Control/Test
Started | 21 | 20
Completed | 21 | 20
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Test/Control | Control/Test
Started | 21 | 20
Completed | 20 | 20
Not Completed | 1 | 0
Not completed — Subject no longer meets the eligibility criteria | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects dispensed a study lens.
Groups:
- All Subjects: All subjects dispensed a study lens.
Arm/Group | All Subjects
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.2 (6.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 39
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: Participants]
  USA | 41

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Lens Centration
Description: Lens centration was assessed using a biomicroscope and was graded using the scale (Grade: 0, 1,2) with grade 0 represent Centered, Grade 1 = Slightly Decentered and Grade 2= substantially decentered. The data was then dichotomized into two groups: those with grade 1 or higher and those with grade 0 (centered). The percentage of participants with Grade 0 Lens centration was reported.
Time Frame: 6 to 8 days
Population: All subjects dispensed at least one study lens.
Measure: Number; unit: Percentage of participants
Groups:
- Test: Subjects that wore the Test lens in either the first or second period of the study.
- Control: Subjects that wore the Control lens in either the first or second period of the study.
Arm/Group | Test | Control
Number analyzed (Participants) | 41 | 41
Percentage of participants | 97.3 | 91.9
Statistical Analysis 1: Comparison: Test vs Control; The proportion of response ("1") was analyzed using a generalized linear mixed model with a binary distribution and logit link function for all questions; Test type: Non-Inferiority — Non-inferiority will be concluded if the lower limit is above 0.67. Superiority will be concluded if the lower limit is above 1.0; Generalized Linear Mixed Model Analysis; Finite-sample corrected Akaike's Information Criterion; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.33 to 6.85] — Odds ratio was calculated as Test/Control

2. Primary Outcome: Percentage of Participants With Lens Movement
Description: Lens movement in primary gaze was assessed using a biomicroscope and was graded using the scale (Insufficient/Unacceptable (-2), Minimal/Acceptable (-1), Optimal (0), Moderate/Acceptable (+1) and Excessive/Unacceptable (+2)) with Optimal (0) representing no lens movement. The data was then dichotomized into two groups: those with Optimal Lens movement and otherwise (-2, -1, +1 and +2). The percentage of participants with Optimal Lens movement was reported.
Time Frame: 6 to 8 days
Population: All subjects dispensed at least one study lens.
Measure: Number; unit: Percentage of participants
Arm/Group | Test | Control
Number analyzed (Participants) | 41 | 41
Percentage of participants | 97.3 | 91.9
Statistical Analysis 1: Comparison: Test vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Generalized Linear Mixed Model Analysis; Finite-sample corrected Akaike's Information Criterion; Odds Ratio (OR) = 0.34, 95% CI 2-sided [0.10 to 1.19] — Odds ratio was calculated as Test over Control

3. Secondary Outcome: Overall Handling Scores
Description: Overall handling was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, aged 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: 6 to 8 days
Population: All subjects who had successfully completed all visits and did not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock. Here 'N' (number of participants analyzed) included all participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: CLUE points
Arm/Group | Test | Control
Number analyzed (Participants) | 37 | 37
CLUE points | 60.3 (19.02) | 55.3 (18.71)
Statistical Analysis 1: Comparison: Test vs Control; Test type: Non-Inferiority — The non-inferiority of the Test lens relative to the Control will be concluded if the lower confidence limit of LSM difference is above the non-inferiority margin -5; Mixed Model Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least square mean difference = -5.98, 95% CI 2-sided [-12.48 to 0.52], Standard Error of Mean 3.202 — Mean difference was calculated as Test minus Control

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 2 weeks per subject
Description: All subjects dispensed at least 1 study lens.
Arm/Group | Test | Control
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 0/41 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT04093258/Prot_SAP_000.pdf